CLINICAL TRIAL: NCT03765736
Title: COLOMATE: Colorectal Cancer Liquid Biopsy Screening Protocol for Molecularly Assigned Therapy
Brief Title: Genetic Testing in Screening Patients With Metastatic or Unresectable Colon or Rectal Cancer for a COLOMATE Trial
Status: Terminated | Type: Observational
Why Stopped: Low accrual
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACCRU-GI-1611; NCI-2018-02862 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-GI-1611 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Results first posted 2024-01-23 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Colon Adenocarcinoma; Metastatic Rectal Adenocarcinoma; Stage III Colon Cancer AJCC v8; Stage III Rectal Cancer AJCC v8; Stage IIIA Colon Cancer AJCC v8; Stage IIIA Rectal Cancer AJCC v8; Stage IIIB Colon Cancer AJCC v8; Stage IIIB Rectal Cancer AJCC v8; Stage IIIC Colon Cancer AJCC v8; Stage IIIC Rectal Cancer AJCC v8; Stage IV Colon Cancer AJCC v8; Stage IV Rectal Cancer AJCC v8; Stage IVA Colon Cancer AJCC v8; Stage IVA Rectal Cancer AJCC v8; Stage IVB Colon Cancer AJCC v8; Stage IVB Rectal Cancer AJCC v8; Stage IVC Colon Cancer AJCC v8; Stage IVC Rectal Cancer AJCC v8; Unresectable Colon Adenocarcinoma; Unresectable Rectal Adenocarcinoma
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (1):
- Screening (genetic testing): Patients submit blood samples for genetic testing.
  Interventions: Other: Genetic Testing

INTERVENTIONS:
Other: Genetic Testing — Undergo genetic testing
  Other Names: genetic analysis; Genetic Examination; Genetic Test

SUMMARY:
This trial screens patients with colon or rectal cancer that has spread to other places in the body (metastatic) or cannot be removed by surgery (unresectable) for genetic mutations for recommendation to a molecularly assigned therapy. Identifying gene mutations may help patients enroll onto target companion trials that target these mutations.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To perform blood-based genomic profiling on patients with treatment refractory metastatic colorectal cancer (CRC) to facilitate accrual to molecularly assigned therapies.

II. To facilitate clinically annotated genomic analyses.

OUTLINE:

Patients submit blood samples for genetic testing.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of adenocarcinoma of the colon or rectum that is metastatic and/ or unresectable
* Progression, intolerance, or contraindication to a fluoropyrimidine (e.g., 5- fluorouracil or capecitabine), oxaliplatin, irinotecan, an anti-VEGF monoclonal antibody (bevacizumab, ziv-aflibercept, or ramucirumab), and an anti-PD-1 monoclonal antibody (nivolumab or pembrolizumab) if tumor has deficient mismatch repair proteins (dMMR) or is microsatellite instability-high (MSI-H)
* For patients with KRAS and NRAS wild-type tumors, progression, intolerance, or contraindication to an anti-EGFR monoclonal antibody (cetuximab or panitumumab)

  * Note: If tissue is known to be positive for HER2 expression (IHC 3+) or the tumor has ERBB2 (HER2) amplification detected by a Clinical Laboratory Improvement Act (CLIA)-certified assay, prior treatment with anti-EGFR therapy is not required
* At least one site of disease that is measurable by Response Evaluation Criteria in Solid Tumors (RECIST) criteria (version 1.1) that has not been previously irradiated; if the patient has had previous radiation to the target lesion(s), there must be evidence of progression since the radiation
* Life expectancy >= 3 months per estimation of investigator
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Capable of understanding and complying with the protocol requirements and has signed the informed consent document
* Satisfy at least one of the following two conditions:

  * Willing and able to provide blood sample for screening purposes
  * Guardant 360 testing completed =< 60 days prior to registration

Exclusion Criteria:

* Evidence within the last 3 years of another malignancy which required systemic treatment. EXCEPTIONS: Non-melanotic skin cancer, carcinoma-in-situ of the cervix, or localized prostate cancer with a current PSA of < 1.0mg/dL on 2 successive evaluations, at least 90 days apart, with the most recent evaluation no more than 4 weeks prior to registration
* Unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee
* History of solid organ transplantation
* Pregnant or planning to become pregnant within the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with adenocarcinoma of the colon or rectum that is metastatic and/ or unresectable
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H Strickler, Principal Investigator — Academic and Community Cancer Research United
Locations (18):
- United States (18):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Screening (Genetic Testing)
Started | 197
Completed | 197
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Screening (Genetic Testing)
Number analyzed (Participants) | 197
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 174
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 24
  White | 132
  More than one race | 1
  Unknown or Not Reported | 19
Region of Enrollment [Number; unit: participants]
  United States | 197
Primary Tumor Site [Count of Participants; unit: Participants]
  Left | 146
  Multiple/Other | 11
  Right | 40

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Who Have an Actionable Genomic Profile
Description: This is defined as a patient who received a trial recommendation per the COLOMATE companion trial recommendation form. Will be presented as a point estimate along with a 95% confidence interval (by Wald asymptotic confidence limit).
Time Frame: 6 months
Population: All eligible patients whose genomic profile was available for COLOMATE steering committee review are included in analysis
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Screening (Genetic Testing)
Number analyzed (Participants) | 191
percent of participants | 37.17 [30.32 to 44.03]

2. Primary Outcome: Companion Trial Enrollment
Description: This is defined as a patient who has an actionable genomic profile that enrolls in their recommended companion trial. Will be presented as a point estimate along with a 95% confidence interval (by Wald asymptotic confidence limit).
Time Frame: 3.5 years
Population: All eligible patients who had an actionable genomic profile were included in analysis
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Screening (Genetic Testing)
Number analyzed (Participants) | 71
percent of participants | 26.76 [16.46 to 37.06]

ADVERSE EVENTS:
Description: Adverse events were not collected for this non-interventional trial
Arm/Group | Screening (Genetic Testing)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/36/NCT03765736/Prot_SAP_ICF_000.pdf